CLINICAL TRIAL: NCT05841940
Title: Mass Balance Study of [14C]HLX208 in China Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HLX208-PK-002
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-04

CONDITIONS: Mass Balance Study in Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]HLX208 (Experimental): Single oral dose of 450mg [14C]HLX208 suspension.
  Interventions: Drug: [14C]HLX208

INTERVENTIONS:
Drug: [14C]HLX208 — Carbon-14 labeled HLX208

SUMMARY:
Mass Balance Study of [14C]HLX208 in China Healthy Subjects.

DETAILED DESCRIPTION:
A phase I study to quantify the total mass balance in healthy subjects after a single dose of [14C]HLX208.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between the ages of 18 and 45 years (inclusive).
2. Subjects weighing ≥ 50 kg and Body Mass Index of 18.0 to 32.0 kg/m2.
3. No sperm donation or fertility plan during the study and within 12 months after the end of the study.
4. Subjects who have voluntarily participated in the study and signed the informed consent form with good compliance.

Exclusion Criteria:

1. Known history of drug or food allergy.
2. Known medical history judged by the investigator as not suitable for the study.
3. Has laboratory or physical examination abnormalities during the screening period.
4. Has a positive test for, HBV，HCV，HIV，or syphilis.
5. Has drug abuse history or positive drug abuse test results.
6. Has diseases affecting the absorption, distribution, metabolism, and excretion of oral drugs.
7. Has any other conditions judged by the investigator as not suitable for the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-06-17 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery of total radioactivity in urine and fecal samples. | Up to 336 hours post dose.
  Mass balance recovery of total radioactivity in urine and fecal samples.
Total radioactivity in plasma PK: Cmax | Up to 240 hours post dose.
  Maximum plasma concentration
Total radioactivity in plasma PK: Tmax | Up to 240 hours post dose.
  Time for Cmax
Total radioactivity in plasma PK: AUC0-t | Up to 240 hours post dose.
  Area under the plasma concentration time profile from time 0 to time of the last quantifiable concentration.
Total radioactivity in plasma PK: AUC0-∞ | Up to 240 hours post dose.
  Area under the plasma concentration time profile from time 0 to infinity.
Total rradioactivity in plasma PK: t1/2 | Up to 240 hours post dose.
  Elimination half-life.
Total radioactivity in plasma PK: CL/F | Up to 240 hours post dose.
  Drug clearance.
Total radioactivity in plasma PK: Vz/F | Up to 240 hours post dose.
  Apparent volume of distribution following oral administration.

SECONDARY OUTCOMES:
HLX208 and metabolite PK: Cmax | Up to 240 hours post dose.
  Maximum plasma concentration
HLX208 and metabolite PK: Tmax | Up to 240 hours post dose.
  Time for Cmax
HLX208 and metabolite PK: AUC0-t | Up to 240 hours post dose.
  Area under the plasma concentration time profile from time 0 to time of the last quantifiable concentration.
HLX208 and metabolite PK: AUC0-∞ | Up to 240 hours post dose.
  Area under the plasma concentration time profile from time 0 to infinity.
HLX208 and metabolite PK: t1/2 | Up to 240 hours post dose.
  Elimination half-life.
Adverse events | Screening up to Day 15
  Number of adverse events, which are any untoward medical occurrence regardless of attribution to study drug in a participant who received study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, Dr., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No